CLINICAL TRIAL: NCT03172715
Title: Prosthesis Versus Osteosynthesis in Treatment of Intra-articular Fractures of Proximal Tibia: A Randomized, Controlled, Trial
Brief Title: Prosthesis Versus Osteosynthesis in Proximal Tibia Fractures
Acronym: POSITIF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Finland Hospital District (Other)
Collaborators: Tampere University Hospital (Other); Coxa, Hospital for Joint Replacement (Other); Oulu University Hospital (Other); Turku University Hospital (Other Government); Kuopio University Hospital (Other); Seinajoki Central Hospital (Other); Paijat-Hame Hospital District (Other)
Responsible Party: Principal Investigator, Juha Paloneva, Department head, adjunct professor, Central Finland Hospital District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnro 6U/2017
Record Dates: First submitted 2017-05-22; First posted 2017-06-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Tibial Fractures
Keywords: Open reduction internal fixation; Arthroplasty; Surgery; Randomized controlled trial
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORIF (open reduction-internal fixation) (Active Comparator): Osteosynthesis with locking plate(s) will be performed using medial and/or lateral incision, according to morphology of the fracture. Additional osteosynthesis material will be used when necessary. The articular surface will be reduced and bone transplantation or bone substitute used if required.
  Postoperatively, touch-down weight bearing will be allowed for 6 weeks, followed by 2 weeks of half-weight-bearing period. A walker or wheelchair will be used when necessary.
  Interventions: Procedure: Locking plate
- TKR (total knee replacement) (Experimental): Arthroplasty of the knee will be performed within two weeks after the fracture. Medial parapatellar approach will be used. The minimal possible constraint of the prosthesis (cruciate retaining, posterior cruciate sacrificing or semi-constrained) will be used. A possible insufficient bone stock may be rebuilt with augments. Hinged prosthesis will be used only if stability of the medial collateral ligament is insufficient. A cemented or uncemented tibial stem extender (minimum length 50mm) will be used in all cases. Additional osteosynthesis will be used when necessary. Postoperatively, the patients will be allowed full weight bearing as tolerated.
  Interventions: Procedure: TKR

INTERVENTIONS:
Procedure: Locking plate — Osteosynthesis
  Arms: ORIF (open reduction-internal fixation)
Procedure: TKR — Total knee arthroplasty
  Arms: TKR (total knee replacement)

SUMMARY:
The aim of this study is to compare knee function and pain one year after treatment of intra-articular proximal tibia fracture using either osteosynthesis with a locking plate (ORIF) or primary total knee replacement (TKR) in patients over 65 years of age.

DETAILED DESCRIPTION:
Intra-articular proximal tibial fractures are relatively common in the elderly. They constitute 8% of all fractures in patients over 65 years. Open reduction and internal fixation (ORIF) is the golden standard treatment for these fractures.

The treatment with ORIF is associated with significant co-morbidity due to complicating concomitant factors, such as osteoporosis, poor co-operation, infection and inadequate stability of osteosynthesis. A high failure rate (30-79 %) of fixation of tibia plateau fractures in elderly people has been reported. Most of these fractures occur in elderly persons who are at risk to lose their ability to walk independently, because of partial immobilization is required initially and full weight bearing is not allowed during 6 to 8 weeks after the operation. The risk of post-traumatic osteoarthritis has been reported to be 5.3-times higher than in the normal population even if adequate stability is achieved and other conditions normalized for fracture healing. It has also been reported that total knee replacement (TKR) performed for post-traumatic arthritis after tibial plateau fracture lead to worse outcome compared with TKR due to primary osteoarthritis. In addition, previous operations increase the risk of complications after TKR. The complication rate in secondary TKR has been reported to be over 18 %.

The available data regarding TKR as a primary treatment option for proximal tibial plateau fracture suggest that fast mobilization and return to normal daily activities may be achieved. These data also suggest a low rate of complications. There are no randomized controlled trials comparing the outcomes of the traditional treatment option (open reduction- internal fixation, ORIF) and TKR as primary treatment of these fractures. In this study investigators compare the outcomes of locking plate osteosynthesis and total knee arthroplasty according to Oxford knee score, pain, ability to walk, or quality of life one year after randomization in 98 patients aged over 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute intra-articular proximal tibia fracture with impression of the joint cartilage (Schatzker grades II to VI)
* Impression of tibial plateau min 2 mm
* Intact patellar tendon
* The patient accepts both treatment options (osteosynthesis and arthroplasty)

Exclusion Criteria:

* Not voluntary
* Previous arthroplasty of the knee
* Previous fracture affecting the knee joint
* Inability to co-operate
* Not independent (institutionalized living before fracture)
* Severe osteoarthritis (Kellgren-Lawrence grade 4)
* Open fracture (Gustilo grade 2 or over)
* Progressive metastatic malign disease
* Multiple fractures requiring operative treatment
* Severe soft tissue injury around the knee (Tscherne classification grade 3)
* Avulsion fracture of the patellar tendon or concomitant patellar tendon tear
* Inability to walk before fracture
* Severe medical comorbidities
* Body Mass Index over 40
* Unacceptably high risk of surgery due to severe medical comorbidities
* Significant arterial or nerve trauma
* Severe substance abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-01-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Knee function | 12 months
  Oxford knee score 12 months after randomisation

SECONDARY OUTCOMES:
Change in knee function | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Change in Oxford knee score
Change in pain | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Numeric rating scale (rest, night, exercise)
Change in physical performance | 6 weeks (TKR only), 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Short Physical Performance Battery (SPPB)
Change in quality of life | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Short form-36 (SF-36)
Reoperations | Up to 10 years following randomisation
  Need for revision surgery
Satisfaction | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Satisfaction with knee (Numeric rating scale, range 0 to 10)

OTHER OUTCOMES:
Pain medication | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Pain medication used (pills per day)
Complications | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Any complication following injury or treatment
Medical and social services (quantity) | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Use of medical and social services (quantity)
Medical and social services (costs) | Baseline, 6 weeks, 3 months, 6 months, 12 months, 24 months, 5 years, 10 years
  Costs of medical and social services used

CONTACTS AND LOCATIONS:
Overall Officials: Juha Paloneva, MD, PhD, Principal Investigator — Central Finland Hospital
Locations (8):
- Finland (8):
  - Central Finland Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Coxa Joint Replacement Hospital, Tampere
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Houdek MT, Watts CD, Shannon SF, Wagner ER, Sems SA, Sierra RJ. Posttraumatic Total Knee Arthroplasty Continues to Have Worse Outcome Than Total Knee Arthroplasty for Osteoarthritis. J Arthroplasty. 2016 Jan;31(1):118-23. doi: 10.1016/j.arth.2015.07.022. Epub 2015 Jul 17. PMID 26264176
- [Background] Wasserstein D, Henry P, Paterson JM, Kreder HJ, Jenkinson R. Risk of total knee arthroplasty after operatively treated tibial plateau fracture: a matched-population-based cohort study. J Bone Joint Surg Am. 2014 Jan 15;96(2):144-50. doi: 10.2106/JBJS.L.01691. PMID 24430414
- [Background] Somersalo A, Paloneva J, Kautiainen H, Lonnroos E, Heinanen M, Kiviranta I. Incidence of fractures requiring inpatient care. Acta Orthop. 2014 Sep;85(5):525-30. doi: 10.3109/17453674.2014.908340. Epub 2014 Apr 3. PMID 24694275
- [Background] Malviya A, Reed MR, Partington PF. Acute primary total knee arthroplasty for peri-articular knee fractures in patients over 65 years of age. Injury. 2011 Nov;42(11):1368-71. doi: 10.1016/j.injury.2011.06.198. Epub 2011 Jul 18. PMID 21763651
- [Background] Kini SG, Sathappan SS. Role of navigated total knee arthroplasty for acute tibial fractures in the elderly. Arch Orthop Trauma Surg. 2013 Aug;133(8):1149-54. doi: 10.1007/s00402-013-1792-8. Epub 2013 Jun 16. PMID 23771128
- [Background] Shimizu T, Sawaguchi T, Sakagoshi D, Goshima K, Shigemoto K, Hatsuchi Y. Geriatric tibial plateau fractures: Clinical features and surgical outcomes. J Orthop Sci. 2016 Jan;21(1):68-73. doi: 10.1016/j.jos.2015.09.008. Epub 2015 Dec 6. PMID 26671570
- [Background] Haufe T, Forch S, Muller P, Plath J, Mayr E. The Role of a Primary Arthroplasty in the Treatment of Proximal Tibia Fractures in Orthogeriatric Patients. Biomed Res Int. 2016;2016:6047876. doi: 10.1155/2016/6047876. Epub 2016 Jan 18. PMID 26885510